CLINICAL TRIAL: NCT00774514
Title: The Cardiovascular Effects of Nitrogen Dioxide Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Umeå University (Other)
Responsible Party: Dr Anders Blomberg, Umeå University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: Dnr 08-113M
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2009-04-09 (Estimated); Status verified 2009-04

CONDITIONS: Endothelial Dysfunction
Keywords: Air Pollution; Nitrogen Dioxide; NO2; Endothelial dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Air exposure (Experimental): 1 hour exposure to filtered air during intermittent exercise
  Interventions: Procedure: Forearm Vascular Study
- NO2 exposure (Experimental): 1 hour exposure to nitrogen dioxide at 4ppm during intermittent exercise
  Interventions: Procedure: Forearm Vascular Study

INTERVENTIONS:
Procedure: Forearm Vascular Study — Forearm venous occlusion plethysmography to measure forearm blood flow during intrabrachial infusion of vasodilators Acetylcholine (5-20 mg/min), sodium nitroprusside (2-8 µg/min), bradykinin (100-1000 pmol/min) and verapamil (10-100 µg/min)
  Other Names: ACh; SNP; BK

SUMMARY:
Exposure to air pollution has been linked to increased cardiorespiratory morbidity and mortality. The exact component of air pollution that mediates this effect is unknown, but the link is strongest for fine combustion derived particulate matter derived from traffic sources. It has been demonstrated that inhalation of diesel exhaust impairs vascular vasomotor tone and endogenous fibrinolysis. Recent studies using an inline retrofit particle trap to reduce the particulate component of exhaust have shown that filtering particles leads to a reversal of the endothelial dysfunction seen after diesel exhaust exposure, and have even suggested an augmentation of vascular function. This raises the question of the cardiovascular effects of the gaseous pollutants, the most abundant of which is nitrogen dioxide. In this study we plan to investigate the cardiovascular effects of nitrogen dioxide exposure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers

Exclusion Criteria:

* Current smokers
* Significant occupational exposure to air pollution
* Regular medication use
* Intercurrent illness

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2008-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Forearm blood flow measured by venous occlusion plethysmography in response to intraarterial vasodilators (acetylcholine, sodium nitroprusside, bradykinin and verapamil) | 4-6 hours after exposure

SECONDARY OUTCOMES:
Plasma t-PA concentrations after infusion of bradykinin | During forearm study
Exhaled nitric oxide | 4-6 hours after exposure

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Sandström, MD PhD, Principal Investigator — Umeå University; Anders Blomberg, MD PhD, Principal Investigator — Umeå University
Locations (1):
- Umeå University, Umeå, Sweden